CLINICAL TRIAL: NCT03089073
Title: Non-interventional Study on Safety and Efficacy of Minirin Melt® in Adult Patients With Nocturia
Brief Title: Study of Minirin Melt® in Adult Patients With Nocturia
Status: Terminated | Type: Observational
Why Stopped: Enrollment challenges
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000208
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Desmopressin — 60μg or 120μg once daily at bedtime
  Other Names: Minirin Melt®

SUMMARY:
Observation of safety and efficacy of Minirin Melt® in adult patients with nocturia

ELIGIBILITY:
Inclusion Criteria:

* Adult aged between 19 and 65 years
* Patients having nocturia
* Decision made to prescribe Minirin Melt according to prescription information
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* When patients have habitual or psychogenic polydipsia (resulting in a urine production exceeding 40ml/kg/24hours)
* When patients have a history of known or suspected cardiac insufficiency and other conditions requiring treatment with diuresis
* When patients have moderate and severe renal insufficiency (creatinine clearance below 50ml/min)
* When patients have known hyponatremia
* When patients have secretion Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
* When patients have hypersensitivity to the active substances or to any of the excipients

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients to whom Minirin melt is prescribed as regular treatment is included in accordance with their usual practice and consistent with Korean prescribing information for Minirin melt.
Sampling Method: Non-Probability Sample
Enrollment: 835 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of nocturnal voids | Baseline and treatment-related visits up to 3 months
  Calculated by 72 hour frequency volume chart (FVC)

SECONDARY OUTCOMES:
Reduction from baseline in the mean number of nocturnal voids | Baseline and treatment-related visits up to 3 months
  Assessed as a (50% decrease) or reduction of nocturnal diuresis (>20%)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Daegu Fatima Hospital (there may be other sites in this country), Daegu, South Korea